CLINICAL TRIAL: NCT03771859
Title: An Observational Study in Patients Receiving Adjuvant Nivolumab Therapy for Resected Melanoma
Brief Title: A Study of Patients Receiving Adjuvant Nivolumab Therapy for Melanoma That Has Been Removed
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-8RX
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants who initiate adjuvant treatment with nivolumab

SUMMARY:
An observational study of melanoma participants who are eligible for and who have initiated treatment with adjuvant nivolumab as part of routine clinical practice.

DETAILED DESCRIPTION:
Participants receiving adjuvant nivolumab therapy could be enrolled prospectively and retrospectively.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a primary diagnosis of melanoma with involvement of lymph nodes or metastatic disease who have undergone complete resection and have no evidence of disease.
* Decision to treat with adjuvant nivolumab therapy has already been taken
* At least 18 years of age at the time of treatment decision
* Patients who provide written informed consent to participate in the study (for retrospectively enrolled patients who are deceased at time of study start, a consent waiver will be sought)

Exclusion Criteria:

* Any patient with a diagnosis of persisting advanced melanoma prior to first administration of nivolumab
* Any patient currently enrolled in an interventional clinical trial for his/her melanoma treatment (note: patients who have completed their participation in an interventional trial or who are no longer receiving the study drug and are only followed up for Overall Survival (OS)/ Relapse Free Survival (RFS) can be enrolled. In case of a blinded study, the treatment arm needs to be known).

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with melanoma with involvement of lymph nodes or metastatic disease who have undergone complete resection, and who receive adjuvant nivolumab under real-world conditions in Belgium or Luxembourg. Patients will be enrolled after complete surgical resection and following a screen procedure (according to standard practice) that shows no evidence of disease. Patients currently enrolled in an interventional clinical trial will not be eligible.
Sampling Method: Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
RFS (relapse free survival) | 5 years

SECONDARY OUTCOMES:
DMFS (distant metastasis free survival) | 5 years
OS (overall survival) | 5 years
Distribution of sociodemographic characteristics in participants initiating nivolumab | 5 years
Distribution of clinical characteristics in participants initiating nivolumab | 5 years
Distribution of treatment patterns in participants initiating nivolumab | 5 years
QOL (quality of life) of patients with resected melanoma receiving adjuvant nivolumab therapy by using the EuroQOL-5D (EQ-5D) | 5 years
  The EQ-5D is a standardized 3-level, 5-dimensional multi-attribute utility questionnaire that measures mobility, self-care, usual activities, pain/discomfort and anxiety/depression, where each dimension is rated by individuals as no problems, slight problems, moderate problems, severe problems, and extreme problems.
The European Organization for Research and Treatment of Cancer (EORTC) QLQ C-30 questionnaire | 5 years
  The EORTC-QLQ-C30 questionnaire is a 30-item instrument that comprises 5 functional scales (physical functioning, cognitive functioning, emotional functioning, social functioning and global quality of life) as well as nine symptom scales (fatigue, pain, nausea/vomiting, dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties).
Functional Assessment of Cancer Therapy-Melanoma (FACT-M) questionnaires | 5 years
  The FACT-M is a frequently used melanoma specific questionnaire which has been validated to assess HRQOL for patients with all stages of melanoma. Besides general questions on Physical Well-Being, Social/Family Well-Being, Emotional Well-Being, and Functional Well-Being, it also contains specific questions related to melanoma, including a subscale on the melanoma surgery
Incidence of AE's | 5 years
Incidence of SAE's | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- Belgium (12):
  - Local Institution, Aalst
  - Local Institution, Antwerp
  - Local Institution, Bouge
  - Local Institution, Bruges
  - Local Institution, Brussels
  - Local Institution, Edegem
  - Local Institution, Ghent
  - Local Institution, Hasselt
  - Local Institution, La Louvière
  - Local Institution, Liège
  - Local Institution, Sint-Niklaas
  - Local Institution, Turnhout
- Local Institution, Luxembourg, Luxembourg

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm